CLINICAL TRIAL: NCT06912789
Title: Are Technological Contributions in Behavior Guidance Techniques Superior to Conventional Methods? : Effects on Dental Anxiety and Pain Perception in Pulpotomy Treatment
Brief Title: Technological Contributions to Behavior Guidance Techniques
Acronym: Pediatrics
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2023/244
Record Dates: First submitted 2025-03-26; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Behavior; Child; Dental Anxiety; Mobile Applications; Pain
MeSH Terms: conditions — Behavior; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: tell-show-do application: The treatment procedure and the exact steps will be explained to the child verbally, after which all the tools and equipment required for the treatment will be shown to the child, before the pulpotomy is performed.
- Group 2: tell-show-do with video modeling application: The treatment procedure and the exact steps will be explained to the child with TSD, a 4 min 33 sec behavioral guidance video will be presented to the child (https://youtu.be/ir1cyjqsWq4?si=pn7jPwzcDfuMHcq).
- Group 3: tell-show-do with mobile phone application: The treatment procedure and the exact steps will be explained to the child with tell-show-do and the Roogies application will be presented to the children together. Roogies is a freely available application (https://apps.apple.com/tr/app/roogies/id1542220556?l=tr).

SUMMARY:
This study aims to evaluate the effects of three different behavior guidance methods on children's dental anxiety and pain perception.

DETAILED DESCRIPTION:
This study will include 63 children aged 6-8 years who will require pulpotomy followed by a Class II composite restoration and will be divided into three groups: tell-show-do (TSD; Group 1), TSD with video modeling (Group 2), and TSD with a mobile phone application (Group 3). Systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and hemoglobin oxygen saturation (SPO2) of the participants will be recorded before the procedure, after local anesthesia, after pulpotomy, and at the end of the procedure. Faces Version of the Modified Child Dental Anxiety Scale (MCDAS f), Wong-Baker Faces Pain Rating Scale (WBFPRS), and Face, Legs, Activity, Cry, Consolability (FLACC) pain scales will be applied.

ELIGIBILITY:
Inclusion Criteria:

* the patients had no previous dental treatment,
* were between ages 6 and 8 years, accepted treatment accompanied by parents,
* scored 3 (positive) or 4 (definitely positive) on the Frankl behavior scale,
* had no systemic disease,
* did not need emergency dental treatment, one of the upper molars required pulpotomy followed by a Class II composite restoration,
* had no mental or physical disabilities,
* understood the commands, and whose parents agreed to participate in the study
* signed the consent form.

Exclusion Criteria:

* Patients who did not meet the inclusion criteria included those who needed other asymptomatic root canal treatment other than pulpotomy indication,
* needed restorative treatment due to a history of dental trauma, those who did not want to be included voluntarily,
* who cried during the procedure or left the treatment unfinished,
* who were determined to be negative (2) or definitely negative (1) according to the Frankl behavior assessment scale.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric population
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of this study will be assessed through physiological measurements ( Blood Pressure) | 3 months
  Systolic Blood Pressure (SBP) and diastolic blood pressure (DBP) will be recorded at multiple time points during the procedure: before the procedure, after the administration of local anesthesia, after pulpotomy, and at the end of the procedure.
  Each patient will rest for 15 minutes before BP measurement. Measurements will be taken from the right wrist with the child in an upright position using an automatic wrist blood pressure device (Wohler, Türkiye). Systolic (SBP) and diastolic blood pressure (DBP) values in cm of mercury (cmHg) will be recorded.
The primary outcomes of this study will be assessed through physiological measurements (Heart rate) | 3 months
  Heart rate (HR) will be measured while the child is in a seated position using a finger-type portable pulse oximeter (Oncomed, USA) attached to the child's right finger. HR values on the digital monitor will be measured as beats per minute.
The primary outcomes of this study will be assessed through physiological measurements (hemoglobin oxygen saturation) | 3 months
  Hemoglobin oxygen saturation (SPO2) will be measured while the child is in a seated position using a finger-type portable pulse oximeter (Oncomed, USA) attached to the child's right finger. SPO2 values on the digital monitor will be measured as a percentage.
The primary outcomes of this study will be assessed through psychometric measurements (The Faces Version of the Modified Child Dental Anxiety Scale) | 3 months
  The Faces Version of the Modified Child Dental Anxiety Scale (MCDAS f) will be used to measure the level of anxiety experienced by the children throughout the procedure.
  For this scale, there are five possible responses consisting of smiling or sad faces, appropriate for each answer given by the child. A happy face corresponds to 1 point whereas a very sad face corresponds to 5 points.
  After the dental treatment, the children in all three groups will be asked the questions, after which the scores corresponding to the facial expressions will be chosen by the children and will be recorded by the pediatric dentist. The total score will be calculated as a minimum of 8 and a maximum of 40, with high anxiety being associated with an increasing score.
The primary outcomes of this study will be assessed through evaluation of dental pain perception (The Wong-Baker Faces Pain Rating Scale) | 3 months
  The Wong-Baker Faces Pain Rating Scale (WBFPRS) will be utilized to assess the pain intensity as reported by the children during the dental treatment.
  Wong-Baker Faces Pain Rating Scale (WBFPRS) includes six facial expressions ranging from a smiling face to a crying face.
  These expressions were explained to the children who were asked to choose the face that best reflected the level of pain they felt during treatment. A smiling face was 0 points (no pain) whereas a crying face was 10 points (very severe pain).
  After physiological and psychometric measurements are recorded, the pediatric dentist will use the WBFBS score to evaluate the children's pain perception. The scoring will be recorded by the same pediatric dentist.
  With high dental anxiety associated with an increasing score.
The primary outcomes of this study will be assessed through evaluation of dental pain perception (Face, Legs, Activity, Cry, Consolability) | 3 months
  The Face, Legs, Activity, Cry, Consolability (FLACC) pain scale will be applied to evaluate the child's pain and distress based on observable behavior during the procedure.
  The measurement will be made by evaluating five behavioral categories (i.e., face, legs, activity, crying, and consolability). Each parameter will be scored between 0 and 2, and the total score will range between 0 and 10, where 0 will indicate calm and comfortable, 1-3 will represent mild discomfort, 4-6 will indicate moderate pain, and 7-10 will signify severe discomfort or pain, or both. A score closer to 10 will indicate severe pain, whereas 0 will mean no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Nil Günaçar, Assoc. Prof., Study Chair — Recep Tayyip Erdogan University Faculty of Dentistry
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yazar M, Aydinoglu S, Gunacar DN. Are technological contributions in behavior guidance techniques superior to conventional methods?: Effects on dental anxiety and pain perception. BMC Oral Health. 2025 May 17;25(1):735. doi: 10.1186/s12903-025-06139-3. PMID 40382626